CLINICAL TRIAL: NCT03296267
Title: Translocation of Microorganisms in Duodenal Biopsies of Healthy Volunteers and Patients With Functional Dyspepsia
Brief Title: Influence of Bile Acids on Bacterial Uptake in Functional Dyspepsia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Purpose: Basic Science
Other Study IDs: s56880
Record Dates: First submitted 2017-09-18; First posted 2017-09-28 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-07

CONDITIONS: Functional Dyspepsia
Keywords: bile acid; bacterial uptake

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- gastroduodenoscopy (Other): all participants undergo a gastroduodenoscopy to use the biopsies in an Ussing chamber experiment.
  Interventions: Procedure: Gastroduodenoscopy

INTERVENTIONS:
Procedure: Gastroduodenoscopy — Gastroduodenoscopy with duodenal biospies: A tube is placed via the mouth into the second part of the duodenum. Biopsy forceps is used to take duodenal biopsies.

SUMMARY:
In up to half of patients seen by gastroenterologists, routine examinations fail to find an underlying organic, systemic, or metabolic disease that readily explains the symptoms. These patients are referred to as patients with disorders of gastrointestinal function, of which functional dyspepsia (FD) is one of the most common. Despite intensive research to investigate various pathophysiological mechanisms of this disease, the pathogenesis remains obscure. The investigators recently demonstrated increased duodenal permeability in FD patients, as assessed by mounting routine endoscopic duodenal biopsy specimens into Ussing chambers to measure transepithelial electrical resistance and passage of a paracellular fluorescent probe. Impaired intestinal barrier function can lead to increased uptake of luminal substances which can induce an immunological response in the mucosa. Interestingly, using transmission electron microscopy (TEM) in duodenal biopsies, the investigators recently observed the presence of a yet to be identified microorganism inside the epithelium and the lamina propria of a subset of FD patients (unpublished observations), suggesting increased translocation of microorganisms.

The aim of the project is to investigate whether FD patients display increased translocation of microorganisms in duodenal biopsies. The investigators will also test the effect of bile acid on translocation of microorganisms and therefore include 20 FD patients and 20 age- and gender-matched healthy volunteers in this study.

DETAILED DESCRIPTION:
The participants will be expected on the department endoscopy of the University Hospital Gasthuisberg, Leuven, Belgium. They are asked to fill in a bundle of questionnaires concerning physical complaints, depression, anxiety (disturbances), pain/disease, body/interoceptive awareness, trauma/abuse and personality. Endoscopy will be performed and up to 8 biopsies will be obtained from the duodenum. All endoscopies will be performed by an experienced endoscopist. Biopsies will be mounted in Ussing chambers and the mucosal compartment will be exposed to commercially available fluorescein-conjugated microorganisms. Uptake of microorganisms will be evaluated by analyzing the serosal compartment and by confocal microscopy of the biopsies. These experiments will also be performed in combination with exposure to bile acids separately and jointly, to assess if bacterial translocation can be exacerbated by these endogenous luminal factors individually and synergistically.

ELIGIBILITY:
Inclusion Criteria:

* Three days before the measurement: no smoking and drinking alcohol
* 12 hours before the measurement: no drinking and eating

Exclusion Criteria:

* symptoms or history of gastrointestinal disease
* first degree relatives with celiac disease
* diabetes mellitus
* allergy/atopy (eczema, asthma, allergic rhinoconjunctivitis)
* coagulation disorders/anticoagulant therapy
* first degree relatives with Crohn's disease or type I diabetes mellitus.
* intake of antihistamines, ketotifen, cromoglycate, acetylsalicylates, NSAIDs, anticholinergics, theophylline, β2-agonists, codeine or opioid derivatives for at least 2 weeks prior to the gastroscopy
* Intake of steroid or immunosuppressive drugs in the last 6 months

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2017-01-02 (Actual); Primary Completion 2018-04-27 (Actual); Study Completion 2018-08-27 (Actual)

PRIMARY OUTCOMES:
Bacterial uptake in the duodenal biopsy measured by fluorescent intensity at the basolateral side of the ussing chamber setup. | 120 minutes
  duodenal uptake of fluorescein conjugated microorganisms

SECONDARY OUTCOMES:
duodenal permeability assessed by measuring transepithelial electrical resistance in the Ussing chamber setup | 120 minutes
  transepithelial electrical resistance

CONTACTS AND LOCATIONS:
Overall Officials: Jan Tack, Professor, Principal Investigator — KU Leuven
Locations (1):
- Translational Research center for Gastrointestinal Disorders (TARGID), Leuven, Vlaams-Brabant, Belgium

IPD SHARING:
Plan to Share IPD: No